CLINICAL TRIAL: NCT07217262
Title: An Open, Single-arm, Single-site Study to Evaluate the Proactive Costs of Care (PCOC) Intervention Delivered by a Trained Lay Educator to Test Feasibility With the Goal of Improving Self-efficacy Among Patients With Gynecologic Cancer on Active Therapy and Their Caregivers
Brief Title: Proactive Costs of Care Study
Acronym: PCOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Foundation for Women's Cancers (Unknown)
Responsible Party: Principal Investigator, Margaret Liang, Principal Investigator, Staff Physician OBGYN, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00003960
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Financial Burden; Financial Toxicity; Financial Stress; Financial Navigation; Gynecologic Cancers; Caregiver Burnout
Keywords: Financial Navigation; Financial Toxicity; Financial Distress; Financial Burden; Gynecologic Cancers; Caregiver Burnout
MeSH Terms: conditions — Financial Stress; Caregiver Burden | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient and Caregiver Arm of Proactive Costs of Care Study (Experimental): No comparator group
  Interventions: Behavioral: Educational Intervention

INTERVENTIONS:
Behavioral: Educational Intervention — Participants will receive the Proactive Costs of Care Guide that covers health insurance, employment, and finding personal and community support. They will also receive the Proactive Costs of Care Cost Tracker to help track medical costs. This one-time intervention can be completed in-person, by video, or by phone. A trained lay educator will spend approximately 30 minutes reviewing health insurance and discussing the 2-3 topics most relevant to the participant. All of the materials are available in a paper version or electronic version.

SUMMARY:
The Proactive Costs of Care intervention is an educational intervention designed to help patients deal with the cost of cancer care. The main goal of this trial is to evaluate whether the Proactive Costs of Care intervention can be successfully delivered to cancer patients who are starting a new treatment and their caregivers by looking at how many participants complete the intervention. The other questions the trial aims to answer are whether the intervention can:

* Improve confidence in solving problems related to costs of care
* Reduce distress related to finances

Participants will complete the Proactive Costs of Care intervention, which is an approximately 30-minute one-time session with a lay educator reviewing the Proactive Costs of Care Guide and Cost Tracker. The intervention can be completed in person, by video, and by phone. Participants will also complete two surveys- one to be completed before the intervention and one to be completed 3 months after the intervention.

DETAILED DESCRIPTION:
The Proactive Costs of Care (PCOC) study aims to assess whether the Proactive Costs of Care intervention can be successfully delivered to cancer patients or their caregivers and help them deal with the costs of cancer care. Patients who are over 18 years of age or older, diagnosed with gynecologic cancer (e.g. endometrial/uterine, cervical, ovarian, vulvar cancers), on active systemic therapy within 30 days of enrollment, receiving treatment at Cedars-Sinai Medical Center, and can speak, read, and understand English are eligible to participate. Caregivers of patients who meet the eligibility criteria above are also eligible to participate.

The Proactive Costs of Care Guide and Cost Tracker were developed with the input of patients, caregivers, social workers, nurses, doctors, and other healthcare workers to address financial burden due to the cost of cancer care. The Proactive Costs of Care Guide covers 3 main topics; health insurance, employment, and personal and community support. The Proactive Costs of Care Cost Tracker helps patients or their caregivers track their medical costs. All of the materials are available in a paper version or electronic version.

Participants will complete a baseline survey before the intervention and a follow-up survey 3 months after the intervention. The patient survey will collect demographic information and ask questions about confidence in solving problems, health insurance literacy, financial distress or well-being, and emotional well-being. The caregiver survey will collect demographic information, confidence in solving problems, health insurance literacy, financial distress or well-being, and caregiver strain.

ELIGIBILITY:
Inclusion Criteria for Patient Participants:

* Individuals 18 years old or older are included.
* Individuals diagnosed with gynecologic cancer
* On active systemic therapy within 30 days of enrollment
* Receiving treatment at Cedars-Sinai Medical Center
* Can speak, read, and understand English

Inclusion Criteria for Caregiver Participants:

- Caregivers to patients who satisfy the criteria above

Exclusion Criteria for Patient and Caregiver Participants:

* Any patients whose records are flagged "break the glass" or "research opt out."
* Cannot speak, read, or understand English
* Not willing to participate in the intervention or complete surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Participant Completion Rate of Educational Intervention | From enrollment to 2 months
  The number of participants who completed the intervention divided by the total number of participants who consented to the study

SECONDARY OUTCOMES:
Change in Self-Efficacy using PROMIS Self-Efficacy | From intervention to 3 months
  Scores range from 10-50, with higher scores indicating more self-efficacy
Change in financial distress using InCharge Financial Distress/Financial Well-Being Scale | From intervention to 3 months
  Scores range from 1-10, with higher scores indicating less financial distress

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Liang, MD, MS, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No